CLINICAL TRIAL: NCT06974331
Title: Effect of Multimedia Protocol About Asthma Control on Asthmatic Children's Adaptation in the Era of Climate Changes
Brief Title: Effect of Multimedia Protocol About Asthma Control
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Esraa Elwan Mohammed Hassan, assistant lecturer at Faculty of Nursing Mansoura University, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: bronchial athama
Record Dates: First submitted 2025-04-22; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-04

CONDITIONS: Bronchial Asthma; Childhood Asthma; Climate Change; Multimedia Learning Education
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multimedia Protocol about Asthma Control (Experimental): Multimedia Protocol about Asthma Control on Asthmatic Children's Adaptation in the Era of Climate Changes
  Interventions: Behavioral: Multimedia Protocol about Asthma Control

INTERVENTIONS:
Behavioral: Multimedia Protocol about Asthma Control — Addressing this multifaceted problem is essential for the well-being of individuals and communities worldwide. Therefore, this study aims to evaluate the effect of multimedia protocol about asthma control on asthmatic children's adaptation in the era of climate.

SUMMARY:
This study aims to evaluate the effect of multimedia protocol about asthma control on asthmatic children's adaptation in the era of climate changes.

DETAILED DESCRIPTION:
In fact, asthma has evolved into a global public health crisis affecting millions of people worldwide . It is one of the most prevalent chronic diseases, with a substantial burden on individuals, families, healthcare systems, and societies as a whole . Asthma not only leads to missed school and work but can also result in severe health emergencies and even death, especially in children . This burden is on the rise, with millions already affected and projections of millions more to come . Furthermore, the complex interplay of genetic, environmental, and lifestyle factors contributing to asthma's development adds to the urgency of addressing this issue . Importantly, the impact of global climate change, with its extreme weather events and increased air pollution, poses an additional threat to asthma sufferers, making it imperative to implement climate change and asthma adaptation measures . The problem's significance is compounded by the vulnerability of children to these environmental changes and the need for innovative strategies like educational multimedia to raise awareness and provide effective interventions. Addressing this multifaceted problem is essential for the well-being of individuals and communities worldwide. Therefore, this study aims to evaluate the effect of multimedia protocol about asthma control on asthmatic children's adaptation in the era of climate.

ELIGIBILITY:
Inclusion Criteria:

* Chronic asthmatic children (aged 7-11 years).
* Both urban and rural asthmatic children.
* Children and their mothers who have not received current or prior guidance about asthma control with the repercussions of climate changes.
* Children whose mothers is educated.

Exclusion Criteria:

* - Children with severe or acute asthma attacks as confirmed by a medical practitioner.
* Any child suffering from other chronic disease or disability, as confirmed by a medical practitioner.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Child awareness about their Asthma Control in the Era of Climate Changes | baseline (day one) and 2 months later as a follow up for each child
  Tool I: A Questionnaire Sheet for Asthmatic Children and their Mothers. This tool will be developed by researcher based on the study aim and after reviewing the related literatures. It will consist of four parts as follows Part One: Sociodemographic Characteristics of Children and their Mothers Part Two: The Child's Clinical Data Part Three: Assessment Questionnaire of Children's Knowledge about Climate Change and their Attitudes Towards Environmental Conservation and Mitigating the Effects of those Changes.
  This part aims to evaluate asthmatic children's knowledge about climate change and their attitudes towards environmental conservation and mitigating the effects of those changes Part Four: Assessment Questionnaire of Child Knowledge about Bronchial Asthma and their Behaviors for Adaptation to Asthma with the Repercussions of Climate Change. This part aims to evaluate asthmatic children's knowledge about their bronchial asthma and their adaptation behavior related to their asthma
Childhood asthma control | baseline (day one) and 2 months later as a follow up for each child
  Tool II; Childhood Asthma Control Test (C-ACT) A valid test that consists of seven questions which aims to assess asthma control in children 4-11 years old and the effects of asthma on daily functioning.
Children adaptation for their Asthma in the Era of Climate Changes | 2 months follow up for each child
  Tool III; Asthma Diary Notes Asthma diaries are daily tracking tools that children can use to monitor their symptoms and medication use.
  this tool aims to follow up children and assess their adaptation for their condition

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No